CLINICAL TRIAL: NCT05371964
Title: An Open Label, Phase 1/1b Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of Imetelstat in Combination With Ruxolitinib in Patients With Myelofibrosis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of Imetelstat in Combination With Ruxolitinib in Participants With Myelofibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MYF1001
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — imetelstat; GRN163L peptide; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Imetelstat sodium + Ruxolitinib (Experimental): Participants who have received ruxolitinib orally (PO) as part of standard of care (SOC) for at least 12 weeks prior to Screening will be enrolled. After enrollment, participants will initiate imetelstat sodium therapy. Dose levels of imetelstat sodium may include 4.7, 6, 7.5, 9.4 mg/kg, until a RP2D is established.
  Interventions: Drug: Imetelstat sodium; Drug: Ruxolitinib
- Part 2: Imetelstat sodium + Ruxolitinib (Experimental): Cohort A: Janus Kinase (JAK) inhibitor naive participants will receive initial treatment with ruxolitinib on study for at least 12 weeks, including 4 consecutive weeks at a stable dose, prior to the addition of imetelstat sodium. Participants can begin imetelstat sodium treatment after sponsor review and approval and meet the following requirements: platelet value is ≥75 x 10^9/L for two consecutive measurements, at least 1 week apart, and the participant does not meet criteria for dose delay.
  Note that the study will no longer recruit participants into Cohort A.
  Cohort B: Participants will receive treatment with ruxolitinib for 12 weeks with at least 4 consecutive weeks at a stable dose prior to enrollment and will start combination treatment with imetelstat on study.
  Interventions: Drug: Imetelstat sodium; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Imetelstat sodium — Imetelstat sodium will be administered as intravenous (IV) every 28 days.
  Other Names: GRN163L
Drug: Ruxolitinib — Ruxolitinib will be administered, orally (PO), twice daily (BID) in cohort B as the standard of care per local prescribing guidelines.

SUMMARY:
The purpose of the study is to identify the recommended Part 2 dose (R2PD) of imetelstat sodium in combination with ruxolitinib in participants with myelofibrosis (MF) in Part 1, and to evaluate the safety and preliminary clinical activity of the R2PD of imetelstat sodium in combination with ruxolitinib in participants with MF in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis (PMF) according to the revised World Health Organization (WHO) criteria or post-essential thrombocythemia-MF or post-polycythemia vera according to the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) criteria.
* Dynamic International Prognostic Scoring System (DIPSS) intermediate-1, intermediate-2 or high-risk MF.
* Candidate for ruxolitinib treatment:

  * Part 1 participants: On ruxolitinib treatment for at least 12 weeks with at least 4 consecutive weeks immediately prior to enrollment at a stable dose.
  * Part 2 participants: Candidate for ruxolitinib treatment as assessed by the investigator and has not previously been treated with a JAK inhibitor (Cohort A) OR currently receiving ruxolitinib per standard of care for at least 12 weeks with at least 4 consecutive weeks at a stable dose prior to enrollment (Cohort B). Note that the study will no longer recruit participants into Cohort A.
* Active symptoms of MF on the MFSAF v4.0 demonstrated by:

  * Part 1 participants only: At least 2 symptoms with a score ≥ 1
  * Part 2 participants only: At least 2 symptoms with a score of ≥ 3, or a total score of at least 10.
* Ineligible for or unwilling to undergo hematopoietic stem cell transplant at time of study entry.
* Hematology laboratory test values within protocol defined limits.
* Biochemical laboratory test values within protocol defined limits.
* Eastern Cooperative Oncology Group Performance Status score of 0, 1, or 2.
* Participants should follow protocol defined contraceptives procedures.
* A woman of childbearing potential must have a negative serum or urine pregnancy test at screening.

Exclusion Criteria:

* Peripheral blood blast count of ≥10% or bone marrow blast count of ≥10%.
* Prior treatment with JAK inhibitor (except for participants being dosed optimized on ruxolitinib treatment prior to screening and enrollment in part 1 or Part 2 Cohort B).
* Known allergies, hypersensitivity, or intolerance to imetelstat or ruxolitinib or excipients.
* Prior treatment with imetelstat.
* Major surgery within 28 days prior to enrollment.
* Any investigational drug regardless of class or mechanism of action, hydroxyurea, chemotherapy, (except for ruxolitinib for participants being dose optimized prior to enrollment), immunomodulatory or immunosuppressive therapy, corticosteroids >30 mg/day prednisone or equivalent ≤14 days prior to enrollment.
* Prior history of hematopoietic stem cell transplant.
* Diagnosis or treatment for malignancy other than MF, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥3 years before enrollment.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
* Clinically significant cardiovascular disease.
* Known history of human immunodeficiency virus (HIV) or any uncontrolled active systemic infection requiring IV antibiotics.
* Active systemic hepatitis infection requiring treatment or any known acute or chronic liver disease unless related to MF. Carriers of hepatitis virus are permitted to enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence, Type, and Severity of Adverse Events, Including Dose-limiting Toxicity (DLT) During the DLT Observation Period and/or Study Treatment | 28 days after first dose
Part 2: Number of Participants With Treatment-emergent Adverse Event (AE) | First dose of study treatment until 30 days after the last dose of study treatment (up to approximately 5 years)
  Safety will be assessed based on incidence and severity (according to Common Terminology Criteria for Adverse Events) of treatment emergent adverse events from the first dose of study treatment until 30 days after completion of treatment.
Part 2: Symptom Response Rate at Week 24 | Week 24
  Symptom response rate is defined as percentage of participants with >=50% reduction in the Total Symptom Score (TSS) measured by the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 e-diary at 24 week compared to baseline.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetic Profile of Ruxolitinib (Maximum Observed Plasma Concentration [Cmax] | From first dose of Ruxolitinib treatment up to approximately 5 years
Part 1: Pharmacokinetic Profile of Ruxolitinib Time to Reach Maximum Plasma Concentration [Tmax]) | From first dose of imetelstat treatment up to approximately 5 years
Part 1 and Part 2: Pharmacokinetic Profile of Imetelstat Sodium Maximum Observed Plasma Concentration [Cmax] | From first dose of imetelstat treatment up to approximately 5 years
Part 1 and Part 2: Pharmacokinetic Profile of Imetelstat Time to Reach Maximum Plasma Concentration [Tmax]) | From first dose of imetelstat treatment up to approximately 5 years
Part 1 and Part 2: Percentage of Participants with Anti-imetelstat Antibodies | From first dose of imetelstat treatment up to approximately 5 years
Part 1: Symptom Response at Week 24 | Baseline, Week 24
  Symptom response rate is defined as percentage of participants with >50% reduction in the TSS measured by the MFSAF v4.0 e-diary at 24 week compared to baseline.
Part 1 and Part 2: Absolute Change From Baseline in TSS at Week 24 | Baseline, Week 24
  Absolute change is defined as change in total symptom score from baseline to week 24 as measured by the MFSAF v4.0 e-diary.
Part 1 and Part 2: Average Absolute Change in TSS Over 24 weeks | Baseline, Week 24
  Average absolute change in TSS is defined as change in the average of absolute change in total symptom score from week 1(baseline) to week 24 as measured by the MFSAF v4.0 e-diary.
Part 1 and Part 2: Spleen Response at Week 24 | Week 24
  Spleen response is the proportion of participants who achieve a reduction in spleen volume of ≥35% from baseline confirmed by magnetic resonance imaging (MRI) or computed tomography (CT).
Part 1 and Part 2: Progression Free Survival (PFS) | From start of study treatment date to the disease progression or death (up to approximately 5 years)
  The time interval from start of study treatment date to the first date of disease progression or death from any cause, whichever occurs first.
Part 1 and Part 2: Percentage of Participants With Complete Remission (CR), Partial Remission (PR), Clinical Improvement (CI) Per the Modified 2013 International Working Group - Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Criteria. | From first dose to end of the treatment (up to approximately 5 years)
Part 1 and Part 2: Time to Response | From first dose of study treatment to the earliest date that a response was first documented (Up to approximately 5 years)
  Time to response was defined as the duration from first dose of study treatment to the earliest date that a response is first documented. The response CI/CR/PR was assessed by IWG-MRT criteria.
Part 1 and Part 2: Duration of Response (DOR) Per IWG-MRT Criteria | From time of initial response to PD or death whichever occurs first (up to approximately 5 years)
  DOR measured from time of initial response (CR/PR/CI) until documented PD or death whichever occurs first.
Part 1 and Part 2: Reduction of Bone Marrow Fibrosis | From first dose to end of the treatment (up to approximately 5 years)
  Reduction of bone marrow fibrosis is defined as the percentage of participants with a post-baseline bone marrow fibrosis degree smaller than the baseline fibrosis degree prior to start of subsequent anticancer therapy.
Part 1 and Part 2: Time to Progression to Acute Myeloid Leukemia (AML) | From first dose to end of the treatment (up to approximately 5 years)
  Time to progression to AML, defined as the time interval from the start of study treatment date to the first date of documented progression to AML or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mudge-Riley, DO, Study Director — Geron Corporation
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - City of Hope, Irvine, California
  - University of Miami, Coral Gables, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Texas Oncology, Denison, Texas
  - Texas Oncology, Tyler, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No